CLINICAL TRIAL: NCT04955210
Title: Establishment of a Multi-Center Big Data System for Severe Infection and a Collaborative Network on Sepsis in Chinese Children
Brief Title: A Multi-Center Data System and Collaborative Network in China for Severe Infection and Sepsis Children
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-18
Record Dates: First submitted 2021-03-26; First posted 2021-07-08 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Critical Illness; Severe Sepsis
Keywords: Sepsis; Critical Illness; severe infection
MeSH Terms: conditions — Critical Illness; Sepsis; Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe infection: Children with severe infection in PICU
  Interventions: Other: Not applicable（Cohort study）

INTERVENTIONS:
Other: Not applicable（Cohort study） — This is a prospective observational study and does not include interventions.

SUMMARY:
1. To research the current situation of severe infection in children in China, and to investigate the incidence, prognosis and disease burden of severe infection in children in different regions of China. 2. Establish the risk prediction model and diagnosi model of severe infection in children, and verify the accuracy of the model in multi-center; 3. To study the effectiveness and safety of different treatments in real diagnosis and treatment, and to evaluate the efficacy of subgroups under different ages and high risk factors.

DETAILED DESCRIPTION:
1.Children between 0 and 18 years old. 2.Severe pneumonia and/or sepsis.Patients were included who meet the guidline for diagnosis and treatment of community-acquired pneumonia in Children (2019) issued by the National Health Commission of the people's Republic of China and/or who meet the International Guide to the 2020 campaign to Save sepsis: management of septic shock and sepsis-related organ dysfunction in children. 3.notifiable infectious diseases.4.The researcher believes that he is not suitable to participate in other situations in this study.5.Participants in other clinical trials in the same period.

ELIGIBILITY:
Inclusion Criteria:

1. Children between 0 and 18 years old.
2. Severe pneumonia and/or sepsis.

Exclusion Criteria:

1. notifiable infectious diseases.
2. The researcher believes that he is not suitable to participate in other situations in this study.
3. Participants in other clinical trials in the same period.

Ages: 29 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children hospitalized in PICU of Children's Hospital of Fudan University from April 2021 to April 2025
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
survival rate | within 28 days after they discharged from PICU
  The survival rate of children in 28 days after their discharged from PICU

SECONDARY OUTCOMES:
length of stay in PICU | within 28 days after they discharged from PICU
  Time from PICU admission to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Guoping Lu, Principal Investigator — The Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No